CLINICAL TRIAL: NCT03267030
Title: Single-Arm PharmacoKinetic/PharmacoDynamic and Safety Study of Eryaspase (GRASPA®) for Patients With Hypersensitivity to PEG-Asparaginase, Diagnosed With Ph(-) Acute Lymphoblastic Leukemia
Brief Title: Asparaginase Encapsulated in Erythrocytes for Patients With ALL and Hypersensitivity to PEG-asparaginase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Birgitte Klug Albertsen (Other)
Collaborators: ERYtech Pharma (Industry)
Responsible Party: Sponsor-Investigator, Birgitte Klug Albertsen, MD PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOR-GRASPALL 2016; 2016-004451-70 (EudraCT Number)
Record Dates: First submitted 2017-05-02; First posted 2017-08-30 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Hypersensitivity to PEG-asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — eryaspase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GRASPA (Experimental): GRASPA will replace remaining PEG-asparaginase doses in case of hypersensitivity.
  Interventions: Drug: GRASPA

INTERVENTIONS:
Drug: GRASPA — Administration of 1-7 doses of 150 IU/kg IV infusion. (every 2 weeks for a maximum of 4 doses and every 6 weeks for maximum 3 doses).
  Other Names: Eryaspase

SUMMARY:
Pegylated-asparaginase (PEG-ASP) is an important part of the treatment of childhood acute lymphoblastic leukaemia (ALL). Unfortunately 13% of patients develops allergy and further treatment is impossible. Furthermore, 6% of patients have developed antibodies (silent inactivation) and have no effect of the PEG-ASP treatment. Truncated asparaginase therapy is associated with inferior event-free survival outcomes, in particular relapse in central nervous system (CNS).

Eryaspase is a new formulation of asparaginase encapsulated in erythrocytes. The erythrocyte membrane protects asparaginase against fast degradation and elimination processes. The encapsulation eliminates the direct somatic contact, and it is hypothesized that this provides the potential to prolong the activity of the enzyme and reduce toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 1-45 years at diagnosis of ALL.
2. First line non-high risk ALL patients enrolled in NOPHO ALL2008 or ALLTogether pilot protocols including PEG-ASNase regimen.
3. Documented hypersensitivity reaction to PEG-ASNase with either:

   Clinical allergy to PEG-ASNase (mild/severe). Serum ASNase activity below the lower level of quantification.
4. Karnofsky/Lansky score ≥50.
5. Ability to understand and willingness to sign a written ICF and to comply with the scheduled visits, treatment plans, laboratory tests and other study procedures. For patients under 18 years of age, either both parents or the legally appointed representatives had to provide consent.

Exclusion Criteria:

1. Philadelphia chromosome positive ALL.
2. Participation in another clinical trial interfering with the study therapy with exception of NOPHO ALL-2008 or ALLTogether pilot protocol. Patients can participate in other clinical trials not interfering with the study drug. In case of doubt this is assessed by the PI.
3. Uncontrolled intercurrent illness including, but not limited to, patients receiving combination antiretroviral therapy or patients with severe or systemic infection, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Other severe acute/chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
5. Pregnant or lactating females (serum human chorionic gonadotropin pregnancy test at screening). Use of a highly effective contraceptive measure in women of child-bearing potential and sexually active girls that are of child-bearing potential is required (contraceptive measures are specified in section 6.0).
6. Inadequate organ functions, which prohibit further asparaginase administration;

   1. History of pancreatitis
   2. History of serious hemorrhage or serious thrombosis with prior asparaginase therapy
   3. Severe hepatic impairment at the time of administration (bilirubin >3 times ULN, transaminases >10 times ULN)
   4. Pre-existing known coagulopathy (e.g. haemophilia)
7. History of grade 3 or higher transfusion reactions or any contraindication to receive blood transfusion. Presence of specific anti-erythrocytes antibodies (auto-antibodies or anti-public antibodies) preventing from getting a compatible packed Red Blood Cells for the patient.
8. Patient under concomitant treatment likely to cause hemolysis.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Klug Albertsen, MD, PhD, Principal Investigator — Pediatric and adolescent medicine, Aarhus University Hospital, Denmark
Locations (23):
- Denmark (6):
  - Aahus University hospial, hematological department, Aarhus, Aarhus C
  - Aarhus University hospital, Aarhus, Aarhus N
  - Aalborg University Hospital, pediatric department, Aalborg
  - Rigshospitalet, Hematological department, Copenhagen
  - Rigshospitalet, Child and Adolescent Medicine, Copenhagen
  - Odense University hospital, pediatric department, Odense
- Estonia (2):
  - Tallin Childrens Hospital, Tallinn
  - Tartu University Clinics, Tartu
- Finland (5):
  - Childrens Hospital, Helsinki. University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - University Hospital of Oulu, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Vilnius University Children's Hospital, Vilnius, Lithuania
- Norway (3):
  - Helse Bergen, Bergen
  - Oslo Universitetssykehus, Rikshospitalet, Oslo
  - St Olavs Hospital, Trondheim
- Sweden (6):
  - Drottning Silvias Barn- och ungdomssjukhus, Gothenburg
  - Universitetssjukhuset Linköping, Linköping
  - Skånes Universitets sjukhus, Lund
  - Astrid Lindgrens Barnsjukhus Karolinska, Stockholm
  - arn- och Ungdomscentrum Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset Uppsala, Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- GRASPA: GRASPA will replace remaining PEG-asparaginase doses in case of hypersensitivity.
  GRASPA: Administration of 1-7 doses of 150 U/kg IV infusion. (For patients coming from NOPHO 2008 (NCT: NCT00819351), eryaspase was administered every 2 weeks for a maximum of 4 doses and every 6 weeks for maximum 3 doses, for patients in the ALLTogether pilot protocol (NCT: NCT03911128) eryaspase was administered at a dose of 150 U/kg every 2 weeks for a maximum of 7 doses).
Period: Overall Study
Arm/Group | GRASPA
Started | 55
Completed | 50
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- GRASPA: GRASPA will replace remaining PEG-asparaginase doses in case of hypersensitivity.
  GRASPA: Administration of 1-7 doses of 150 U/kg IV infusion. (For patients coming from NOPHO 2008, eryaspase was administered every 2 weeks for a maximum of 4 doses and every 6 weeks for maximum 3 doses, for patients in the ALLTogether pilot protocol eryaspase was administered at a dose of 150 U/kg every 2 weeks for a maximum of 7 doses).
Arm/Group | GRASPA
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.1 [3.5 to 10.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 15
  Norway | 5
  Finland | 8
  Denmark | 10
  Lithuania | 14
  Estonia | 3

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics ASNase Activity >100 U/L at 14 Days
Description: The primary endpoint was the percentage of patients with ASNase activity >100 U/L at 14 days following the first infusion (nadir). ASNase activity >100 U/L is considered adequate for complete asparagine depletion in the blood.
Time Frame: 14 days after first infusion
Population: The primary Evaluable Patients (EP) Population was used for the analysis of the primary and key secondary endpoints, defined as all patients recruited into the study who provided data on ASNase level on Day 14 (±2 days) following the first administration of eryaspase.
  All included patients (55) completed first infusion, only in 53 patients an ASNase activity measurement was available.
Measure: Number; unit: percentage of patients
Arm/Group | GRASPA
Number analyzed (Participants) | 53
percentage of patients | 92.5

2. Secondary Outcome: Pharmacokinetic Parameters
Description: Percentage of patients with ASNase activity >100 U/L at 14 days following the fourth infusion of the 2-week dosing intervals. ASNase activity >100 U/L is considered adequate for complete asparagine depletion in the blood.
Time Frame: 14 days after fourth infusion
Population: A total of 12 patients completed 4 infusions with a 2-week interval of these 9 patients had an ASNase activity measurement 14 days following the fourth infusion.
Measure: Number; unit: percentage of patients
Arm/Group | GRASPA
Number analyzed (Participants) | 9
percentage of patients | 66.7

ADVERSE EVENTS:
Time Frame: From first study drug administration and until 30 days after last administration, up to 1 year
Groups:
- Intervention: GRASPA will replace remaining PEG-asparaginase doses in case of hypersensitivity.
  GRASPA: Administration of 1-7 doses of 150 U/kg IV infusion. (For patients coming from NOPHO 2008, eryaspase was administered every 2 weeks for a maximum of 4 doses and every 6 weeks for maximum 3 doses, for patients in the ALLTogether pilot protocol eryaspase was administered at a dose of 150 U/kg every 2 weeks for a maximum of 7 doses).
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 1/55
Serious Adverse Events (participants affected / at risk) | 6/55
Other Adverse Events (participants affected / at risk) | 18/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=55)
hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1)
Hypersenditivity (Immune system disorders) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=55)
Constipation (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (9)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Alanine aminotransferase increase (Investigations) | 1 (1)
hyperlipidemia (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Hypersensibility (Immune system disorders) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1)
Febrile Neutropenia (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
hyperthermia (General disorders) | 1 (1)
rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03267030/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT03267030/SAP_001.pdf